CLINICAL TRIAL: NCT04625569
Title: Role of Genetic Determinants in the Response to Acute Saline Load Testing in Patients With Essential Hypertension (Naload)
Brief Title: Genetic of Response to Acute Saline Load Test in Hypertension (Naload)
Acronym: Naload
Status: Recruiting | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Chiara Lanzani, Medical doctor in nephrology unit, nephrologist, Ospedale San Raffaele
Other Study IDs: Naload
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Hypertension,Essential; Salt; Excess; Genetic Hypertension; Genetic Predisposition to Disease
Keywords: hypertension; salt sensitivity; genetic
MeSH Terms: conditions — Essential Hypertension; Genetic Predisposition to Disease; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and urinary sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NHP referred to our outpatient clinic will be enrolled (150 newly recruited) in acute saline test for phenotype characterisation of PNat relationship(7). For each patient we will collect urine and blood samples for standard clinical biochemistry, including electrolytes, creatinine, EO, aldosterone, plasma renin activity, urinary uromodulin (ELISA), urinary and serum uric acid and blood samples for genetic test.

DETAILED DESCRIPTION:
Acute salt load test: after the equilibration period and achievement of a steady state, a constant-rate i.v. infusion of 2 L of 0.9% NaCl was carried out in 2 hours. BP (mean of 3 measurements taken 3 minutes apart) was measured every 30 minutes during the 2 hours of loading and 3 times at 3-min intervals at the end of the infusion. These last 3 BP values were averaged and used in the analysis.

The results of these tests will be added to an already collected database of salt load test collected in the previous studies (already published)

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65years;
* body mass index (BMI) <30 kg/m2;
* Na intake, evaluated as urinary Na excretion of <300 mEq/24 hours; .office systolic BP (SBP) >140 mm Hg and diastolic BP (DBP) >90 mm Hg in 3 consecutive visits to their family doctors.

Exclusion criteria:

* Female patients
* history of myocardial infarction,
* stroke,
* congestive heart failure,
* liver disease, secondary cause of hypertension,
* diabetes,
* severe hypertension (>160/110 mm Hg),
* abuse of drugs or alcohol, .creatinine clearance < 80 mL/m.

Secondary forms of hypertension (e.g. primary aldosteronism) were ruled out with specific investigations when deemed appropriate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enrolled newly discovered, never treated, mild hypertensive male patients in the 'Outpatient Clinic for Hypertension' of San Raffaele Hospital, Milan (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
DMBP120 | 120 min
  Blood pressure variation at the end of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Lanzani, Doctor, Principal Investigator — Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Trudu M, Janas S, Lanzani C, Debaix H, Schaeffer C, Ikehata M, Citterio L, Demaretz S, Trevisani F, Ristagno G, Glaudemans B, Laghmani K, Dell'Antonio G; SKIPOGH team; Loffing J, Rastaldi MP, Manunta P, Devuyst O, Rampoldi L. Common noncoding UMOD gene variants induce salt-sensitive hypertension and kidney damage by increasing uromodulin expression. Nat Med. 2013 Dec;19(12):1655-60. doi: 10.1038/nm.3384. Epub 2013 Nov 3. PMID 24185693
- [Background] Citterio L, Delli Carpini S, Lupoli S, Brioni E, Simonini M, Fontana S, Zagato L, Messaggio E, Barlassina C, Cusi D, Manunta P, Lanzani C. Klotho Gene in Human Salt-Sensitive Hypertension. Clin J Am Soc Nephrol. 2020 Mar 6;15(3):375-383. doi: 10.2215/CJN.08620719. Epub 2020 Jan 28. PMID 31992575
- [Background] Lanzani C, Gatti G, Citterio L, Messaggio E, Delli Carpini S, Simonini M, Casamassima N, Zagato L, Brioni E, Hamlyn JM, Manunta P. Lanosterol Synthase Gene Polymorphisms and Changes in Endogenous Ouabain in the Response to Low Sodium Intake. Hypertension. 2016 Feb;67(2):342-8. doi: 10.1161/HYPERTENSIONAHA.115.06415. Epub 2015 Dec 14. PMID 26667413
- [Background] Citterio L, Ferrandi M, Delli Carpini S, Simonini M, Kuznetsova T, Molinari I, Dell' Antonio G, Lanzani C, Merlino L, Brioni E, Staessen JA, Bianchi G, Manunta P. cGMP-dependent protein kinase 1 polymorphisms underlie renal sodium handling impairment. Hypertension. 2013 Dec;62(6):1027-33. doi: 10.1161/HYPERTENSIONAHA.113.01628. Epub 2013 Sep 23. PMID 24060892